CLINICAL TRIAL: NCT00528710
Title: Double-Blind, Placebo-Controlled Trial of the Impact of S-Adenosyl-L-Methionine (SAM-e) on the Mood and Other Symptoms in Fibromyalgia
Brief Title: Efficacy of S-Adenosylmethionine in Fibromyalgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Deakin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DUHREC06
Record Dates: First submitted 2007-09-11; First posted 2007-09-12 (Estimated); Last update posted 2007-09-12 (Estimated); Status verified 2007-09

CONDITIONS: Fibromyalgia Syndrome
Keywords: S-Adenosylmethionine
MeSH Terms: conditions — Fibromyalgia | interventions — S-Adenosylmethionine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- P (Placebo Comparator): Placebo Control Group
  Interventions: Dietary Supplement: SAM-e (S-Adenosyl-L-Methionine)

INTERVENTIONS:
Dietary Supplement: SAM-e (S-Adenosyl-L-Methionine) — One 400 mg tablet daily in the morning.

SUMMARY:
Fundamentally, the trial aims to conduct a gold-standard test of the clinical impact of SAM-e in the treatment of depressed mood and general symptoms of fibromyalgia (FMS).

As such, salient clinical and pathological parameters will be assessed over an 8-week period in 60 patients who will be provided with either SAM-e or a placebo preparation . On the basis of previous literature, it is hypothesised that patients in the active treatment group will experience moderate but significant improvements across the clinical measures, and that these gains will be significantly greater than any reported in the placebo group. All patients will provide informed consent. All procedures will be conducted under medical supervision and the preparation itself is very safe when used in the manner proposed for the trial

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Fibromyalgia by a medical practitioner

Exclusion Criteria:

* Pregnancy, Manic and hypomanic conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2006-11; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Symptom reduction in Fibromyalgia. Specifically we expect a reduction in depressive symptoms, sleep disturbances and gastric disturbances. | Measured at three points in time: pre-trial and at 4 and 8 weeks

SECONDARY OUTCOMES:
Examination of dose-response data and the nature of the placebo effect in these conditions. | Measured at three points in time: pre-trial and at 4 and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Tooley, PhD, Principal Investigator — Deakin University
Locations (1):
- Deakin University, Burwood, Victoria, Australia